CLINICAL TRIAL: NCT02959671
Title: Clinical Performance of a New Esthetic, Self-ligating Orthodontic Bracket
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: 3M Oral Care (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1611M00321
Record Dates: First submitted 2016-11-02; First posted 2016-11-09 (Estimated); Results first posted 2021-01-14 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2020-12

CONDITIONS: Malocclusion
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lower Anterior EXD-952 Self-ligating Brackets (Experimental)
  Interventions: Device: Lower Anterior EXD-952 Self-ligating Brackets

INTERVENTIONS:
Device: Lower Anterior EXD-952 Self-ligating Brackets — Placement of EXD-952 Self-ligating Brackets on mandibular incisors

SUMMARY:
A cohort of 15 patients starting orthodontic treatment with fixed appliances will receive EXD-952 Ceramic Self-ligating brackets on all mandibular incisors and a different type of brackets on the remaining mandibular teeth. Tooth movement will be initiated using 0.014" or 0.016" Nickel-Titanium archwires.

A second cohort of 15 patients will receive EXD-952 Ceramic Self-ligating bracket on all mandibular incisors in a later phase of their ongoing orthodontic treatment. The mandibular incisor brackets will be removed and EXD-952 Ceramic Self-ligating brackets placed instead. Other mandibular brackets will remain in place. Tooth movement will be performed using 0.019x0.025" Stainless Steel archwires.

In both cohorts bracket door stability, the ability of the door to hold the archwire in the bracket slot, the bracket's ability to rotate teeth, clinicians' satisfaction with the bracket, and patient comfort in comparison with other brackets will be assessed.

The evaluation for each patient will last for at least until one archwire change (cohort 1) or one appointment interval (6-8 weeks, cohort 2).

After the evaluation period, EXD-952 Ceramic Self-ligating brackets will remain in place until the orthodontic treatment is completed.

ELIGIBILITY:
Inclusion Criteria:

* Permanent mandibular dentition including incisors, canines, premolars, and first molars (includes subjects treated with the extraction of premolars)
* Mandibular incisors with sound, non-carious buccal enamel and no pretreatment with chemical agents such as hydrogen peroxide

Exclusion Criteria:

* Mental/emotional/developmental disability
* Inability to give informed consent
* Cleft lip and/or palate, craniofacial anomaly, or syndrome
* Obvious oral hygiene issues such as excessive plaque accumulation, gingivitis, and/or pre-existing white spot lesions
* Prosthodontic or restored substrate extending on the labial surface of mandibular incisors
* Deep bite
* Known allergies to any study materials

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-01; Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lower Anterior EXD-952 Self-ligating Brackets
Started | 34
Completed | 29
Not Completed | 5
Not completed — Adverse Event | 2
Not completed — Participants signed a consent; however enrollment was complete before they started study activity. | 3

BASELINE CHARACTERISTICS:
Population: Baseline data was collected from 31 patients out of the 34 who signed the consent. Three participants signed the consent, but did not participate in data collection. They are excluded from baseline analysis.
Arm/Group | Lower Anterior EXD-952 Self-ligating Brackets
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.8 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 31
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Bracket Door Stability
Description: The stability of the bracket door is assessed at the time of bracket placement. Each bracket has 4 doors. Outcome is reported as the percent of bracket doors across all participants that break at bracket placement. Number of total broken bracket doors/number of total bracket doors across all participants * 100. Unit of measure is "percentage of bracket doors."
Time Frame: baseline
Population: All participants who participated in data collection for this measure are included.
Measure: Number; unit: percentage of bracket doors
Arm/Group | Lower Anterior EXD-952 Self-ligating Brackets
Number analyzed (Participants) | 31
percentage of bracket doors | 0.8

2. Primary Outcome: Ability of Door to Successfully Hold the Archwire in the Bracket Slot
Description: The ability of door to hold the archwire in the bracket slot is assessed at the time of bracket placement. If the door is unable to hold the archwire, then spontaneous door opening occurs. Each bracket has 4 doors. Outcome is reported as the percent of bracket doors that successfully held the archwire within the bracket slot at bracket placement. Number of successful bracket doors/number of total bracket doors across all participants * 100. Unit of measure is "percentage of bracket doors."
Time Frame: baseline
Population: All participants who participated in data collection for this measure are included.
Measure: Number; unit: percentage of bracket doors
Arm/Group | Lower Anterior EXD-952 Self-ligating Brackets
Number analyzed (Participants) | 31
percentage of bracket doors | 96

3. Primary Outcome: Bracket's Ability to Rotate Teeth
Description: The bracket's ability to rotate teeth will be assessed after the first archwire change (expected 6-8 weeks after initial bonding). Clinician will rate rotational correction as adequate or not adequate. Outcome is reported as the percent of participants for whom the clinician rated rotational correction as adequate.
Time Frame: 6-8 weeks
Population: All participants who participated in data collection for this measure are included.
Measure: Number; unit: percent of participants
Arm/Group | Lower Anterior EXD-952 Self-ligating Brackets
Number analyzed (Participants) | 31
percent of participants | 62.5

4. Primary Outcome: Clinicians' Satisfaction With the Bracket
Description: The clinician's satisfaction with the bracket will be assessed after the first archwire change (expected 6-8 weeks after initial bonding). Clinician will rate their satisfaction on a 5-point Likert scale (Very unsatisfied, somewhat unsatisfied, neutral, somewhat satisfied, very satisfied). A rating of 4 (somewhat satisfied) or 5 (very satisfied) is considered successful. Outcome is reported as the percent of participants for whom the clinician rated bracket satisfaction as somewhat satisfied or very satisfied.
Time Frame: 6-8 weeks
Population: All participants who participated in data collection for this measure are included.
Measure: Number; unit: percent of participants
Arm/Group | Lower Anterior EXD-952 Self-ligating Brackets
Number analyzed (Participants) | 31
percent of participants | 70

5. Primary Outcome: Patient Comfort in Comparison With Other Brackets (Questionnaire)
Description: The patient's comfort in comparison with other brackets will be assessed after the first archwire change (expected 6-8 weeks after initial bonding). Patients will rate their satisfaction on a 5-point Likert scale (Very unsatisfied, somewhat unsatisfied, neutral, somewhat satisfied, very satisfied). A rating of 4 (somewhat satisfied) or 5 (very satisfied) is considered successful. Outcome is reported as the percent of participants who rated their comfort in comparison with other brackets as somewhat satisfied or very satisfied.
Time Frame: 6-8 weeks
Population: All participants who participated in data collection for this measure are included.
Measure: Number; unit: percent of participants
Arm/Group | Lower Anterior EXD-952 Self-ligating Brackets
Number analyzed (Participants) | 31
percent of participants | 84

ADVERSE EVENTS:
Time Frame: at least 6 weeks
Groups:
- Lower Anterior EXD-952 Self-ligating Brackets: Adverse event data was collected from 31 patients out of the 34 who signed the consent. Three participants signed the consent, but did not participate in data collection. They are excluded from data analysis.
Arm/Group | Lower Anterior EXD-952 Self-ligating Brackets
All-Cause Mortality (participants affected / at risk) | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 2/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lower Anterior EXD-952 Self-ligating Brackets (N=31)
Enamel Wear of the Maxillary Incisors (Product Issues) | 2 (2) — Adverse device effect

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2016-12-20): https://cdn.clinicaltrials.gov/large-docs/71/NCT02959671/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2016-11-03): https://cdn.clinicaltrials.gov/large-docs/71/NCT02959671/Prot_SAP_001.pdf